CLINICAL TRIAL: NCT06367543
Title: Guideline-recommended Basic Parameter Adherence in Neurocritical Care Patients: German-wide Observational Multicenter Individual Participant Data Meta-analysis
Brief Title: Guideline-recommended Basic Parameter Adherence in Neurocritical Care Patients
Acronym: NORMONICU
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: University of Leipzig (Other); University of Wuerzburg (Other); Technical University of Munich (Other); Heidelberg University (Other); University of Cologne (Other); University of Mannheim (Other); University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 117/22
Record Dates: First submitted 2024-03-13; First posted 2024-04-16 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: neurocritical care unit; guideline adherence; stroke; intracerebral hemorrhage; ischemic stroke; targeted management
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Ischemic Stroke | interventions — Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stroke admitted to an NICU: Patients with neurovascular disease necessitating NICU-treatment. Neurovascular disease includes all stroke subcategorized into ischemic stroke and hemorrhagic stroke (i.e. subarachnoid hemorrhage and intracerebral hemorrhage)
  Interventions: Diagnostic Test: Time in therapeutic range of vital parameters

INTERVENTIONS:
Diagnostic Test: Time in therapeutic range of vital parameters — Treatment adherence on NICU to the following vital parameters:
  1. Temperature (T<37,5°C) (every 4 hours during the first 96 h after admission to neurocritical care unit)
  2. systolic blood pressure ICD-10 (International Statistical Classification of Diseases 10th Revision) (I60, 161 & 162): 100-140 mmHg ICD-10 (I63): 120-180 mmHg (every 4 hours during the first 96 h after admission to neurocritical care unit)
  3. Mean arterial blood pressure (MAP: 60-90 mmHg) (every 4 hours during the first 96 h after admission to neurocritical care unit)
  4. Arterial oxygen partial pressure (paO2: 75 - 100 mmHg) (every 4 hours during the first 96 h after admission to neurocritical care unit)
  5. Arterial carbon dioxide partial pressure (paCO2: 35 - 45 mmHg). (every 4 hours during the first 96 h after admission to neurocritical care unit)
  6. Blood glucose (BG: 80-180 mg/dL). (every 4 hours during the first 96 h after admission to neurocritical care unit)
  Other Names: Treatment adherence on NICU

SUMMARY:
The aim of the planned study project is to assess the current situation regarding the treatment of patients with severe stroke at the neuro-critical care unit. Specifically, determination of whether the target parameters recommended in the guidelines for temperature, systolic blood pressure, mean arterial blood pressure, blood glucose, arterial oxygen partial pressure and arterial carbon dioxide partial pressure had to be maintained. From the planned data analysis, the need for the introduction of cerebrovascular bundles can be derived and planned.

DETAILED DESCRIPTION:
Cerebrovascular events include cerebral infarctions as well as intracranial haemorrhages. If the severity of this cerebrovascular damage is so severe, functional damage to the brain occurs, which must be treated regularly in intensive care. In particularly severe cases, patients are analgosedated, intubated and ventilated to treat elevated intracranial pressure (ICP). Especially in these critically ill patients, it is known from numerous studies that adherence to normal physiological parameters of body temperature, blood pressure, serum glucose and ventilation parameters leads to an improvement in the outcome of the patients. This has led to the corresponding guidelines for the treatment of these patients.

In the case of patients with sepsis, it is known that a scientifically proven finding of a better treatment option did not directly lead to an implementation in daily patient care. Only the introduction of treatment and target bundles as a combination of such interventions then led to the implementation of the recommendations and to an improvement in patient care. From this background, the question arises as to whether the above-mentioned measures have been implemented in neurological intensive care medicine for patients with severe cerebrovascular diseases or whether measures such as the introduction and training of target bundles could be useful.

The aim of this research project is to generate new evidence for or against common treatment algorithms in fields where no randomized data are available. Among other things, it will be analysed to what extent early management on intensive care units affect outcomerelevant parameters. The overall aim is to improve the current level of evidence on the management of patients with severe stroke by analyzing a large database of individualized patient data.

The aim of the planned study project is a national, multicentre retrospective collection of real patient data in specialized neurological/neurosurgical intensive care units of patients with severe cerebrovascular diseases. From these collected data, the reality of treatment is to be presented and guideline adherence is to be calculated. From the planned data analysis, the need for the introduction of cerebrovascular bundles can be derived and planned.

Specifically, a retrospective evaluation of patients who were hospitalized at eight neurocritical care units in eight tertiary centres in Germany. Specifically, it is planned to first identify these patients through a controlling query. Subsequently, various clinical parameters from the routine acute phase will be collected by reviewing the in-house electronic data systems. Aspects of data protection will be observed according to the local institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* acute neurovascular disease, i.e. cerebral ischemia, intracerebral hemorrhage or subarachnoid hemorrhage (International Classification of diseases, ICD10, i.e. 160.x, 161.x, 163.x).
* neurocritical care admission due to intubation and controlled ventilation Stay ≥ 4 days at the ICU.
* Hospital stay on NICU of a minimum of 4 days.

Exclusion Criteria:

Patients who received initial do-not-treat/do-not-resuscitate (DNT/DNR) orders as well as those who deceased within 24 hours after admission were not enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted with the diagnosis of stroke treated on NICU will be included.
Sampling Method: Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time in Therapy range | every 4 hours during the first 96 hours after admission to neurocritical care unit.
  Percentage of patients within treatment range for the primary intervention measured parameters every 4 hours during the first 96 hours after admission to neurocritical care unit:
  * Body temperature < 37,5 degrees celsius.
  * Systolic blood pressure range by patients with ischemic stroke (120-180 mmHg; systolic blood pressure range by patients with hemorrhagic stroke (100-140 mmHg.
  * Mean blood pressure range in all patients (60-90 mmHg).
  * Serum blood glucose range (80-180 mg/dL).
  * Arterial oxygen partial pressure paO2 range (75-100 mmHg)
  * Arterial carbon dioxide partial pressure (paCO2) range (35-45 mmHg).

SECONDARY OUTCOMES:
Acute measures | From date of admission to the neurocritical care unit until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days.
  1. Percentage of participant with preclinical intubation.
  2. Percentage of participants who received intravenous thrombolysis
  3. Percentage of participants who received mechanical thrombectomy with TICI grading (Thrombolysis in cerebral infarction (TICI) scale), (minimum value of 0 and maximum value of 3; higher scores mean better outcome).
  4. Percentage of participants who received Clipping/Coiling during the stay at the neurocritical care unit.
  5. Percentage of participant who received surgical hematoma evacuation during the stay at the neurocritical care unit.
Invasive measures performed in the course of the Stay | From date of admission to the neurocritical care unit until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days.
  1. Active cooling system. (Percentage of participants with active cooling system from the whole study population).
     * Percentage of participants who received invasive (Cooling catheter for temperature management).
     * Percentage of participants who received surface cooling pads.
  2. Percentage of participant with Placement of EVD (External ventricular drain)
  3. Percentage of participants with placement of lumbar drain.
Duration of ventilation | From date of admission to the neurocritical care unit until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days.
  Duration of ventilation measured in hours.
Deceased on Intensive Care. | From date of admission to the neurocritical care unit until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days.
  Death on neurocritical care Unit.
NIHSS (National Institutes of Health Stroke Scale). | From date of admission to the neurocritical care unit until the date of discharge or date of death from any cause, whichever came first, assessed up to 90 days.
  NIHSS (National Institutes of Health Stroke Scale) on discharge or transfer. (minimum value of 0 and maximum value of 42; higher scores mean worse outcome) on discharge or transfer.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Gießen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Mullhi RK, Singh N, Veenith T. Critical care management of the patient with an acute ischaemic stroke. Br J Hosp Med (Lond). 2021 Jan 2;82(1):1-9. doi: 10.12968/hmed.2020.0123. Epub 2021 Jan 18. PMID 33512282
- [Background] Sharma D, Smith M. The intensive care management of acute ischaemic stroke. Curr Opin Crit Care. 2022 Apr 1;28(2):157-165. doi: 10.1097/MCC.0000000000000912. PMID 35034076
- See also: Guidelines of the German Society of Neurology for the acute treatment of ischemic stroke — http://dgn.org/leitlinie/akuttherapie-des-ischamischen-schlaganfalls
- See also: Guidelines of the German Society of Neurology for the treatment of intracerebral hemorrhage — http://dgn.org/leitlinie/behandlung-von-spontanen-intrazerebralen-blutungen